CLINICAL TRIAL: NCT05958316
Title: A Randomized Controlled Trial Using a Heuristic Tool To Improve Symptom Self-Management in Adolescents and Young Adults With Cancer
Brief Title: Heuristic Tool To Improve Symptom Self-Management in Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22-20031; HM20025194 (Other: Virginia Commonwealth University); SSU00210247 (Other: Advarra); 1R01CA286799-01 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Symptoms and Signs; Cancer; Childhood Cancer
Keywords: Supportive Care; Symptom Management
MeSH Terms: conditions — Signs and Symptoms; Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Symptom Assessment Tool C-SCAT (Experimental): Participants will be asked to complete the C-SCAT at three of their clinic visits for cancer treatment in addition to usual care for assessing symptoms. This intervention period will last up to about 12 weeks, depending on cancer treatment schedule (for example, every 2, 3 or 4 weeks).
  Interventions: Behavioral: Computerized Symptom Capture Tool (C-SCAT) Intervention
- Usual Care Control Group (Active Comparator): Participants will follow usual care for cancer symptoms for up to 12 weeks, depending on how cancer treatment schedule (for example, every 2, 3 or 4 weeks).
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Computerized Symptom Capture Tool (C-SCAT) Intervention — The C-SCAT includes the 32 symptoms from the Memorial Symptom Assessment Scale (MSAS). Users select symptoms they have experienced over the past week, rate each symptom's severity and distress, and name a perceived cause. They then identify temporal and causal relationships between symptoms using lines and arrows, designate groups, i.e., "clusters" of symptoms, and give a name to each cluster. They are asked the reason for a symptom's designation as a priority symptom and what they do to alleviate that symptom. Next, they are asked to designate a priority cluster and finally, to confirm whether the image accurately reflects their symptom experience. Then, at the clinic visit, the AYA shares the visual image with the HCP, and more importantly, their priority symptoms, which can facilitate the symptom discussion. The C-SCAT intervention group will complete the C-SCAT prior to each of three encounters with their health care providers (HCPs).
  Arms: Computerized Symptom Assessment Tool C-SCAT
Behavioral: Usual Care Control — Usual care is defined as the usual approach to assessing symptoms during the HCP encounter. To provide attentional control to the usual care control group and prevent disproportionate attrition from that group, study staff will contact participants three times during the intervention period (approximately 3 months) when they are in for a scheduled clinic visit and communicate the following: 1) express appreciation for ongoing study participation; 2) ask how everything is going with their treatment; 3) ask if anything has changed with their treatment plan since the last study visit; and 4) confirm continued participation in the study.
  Arms: Usual Care Control Group

SUMMARY:
Determine the effects of the Computerized Symptom Assessment Tool (C-SCAT) versus usual care on the primary outcomes of self-efficacy for symptom management and symptom self-management behaviors

DETAILED DESCRIPTION:
This is a multi-site two-group randomized control trial (RCT) design to evaluate the effects of the Computerized Symptom Assessment Tool (C-SCAT) for improving symptom self-management versus usual care in 126 adolescents and young adults (AYAs) who are within the first three months of a diagnosis of cancer and who are receiving cancer treatment. For this study, cancer treatment will be defined as a prescribed infusion ( e.g., chemotherapy, immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Has received at least 1 cycle of cancer treatment and is within 3 months of initial cancer diagnosis
* Receiving regularly scheduled cancer treatment and will be receiving at least three more cycles
* Reports at least 1 symptom related to cancer and/or its treatment
* Able to speak, read, and write English as required for completion of the C-SCAT and study measures

Exclusion Criteria:

- Cognitive and/or physical inability to complete study measures.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Effects of the C-SCAT versus usual care on the primary outcomes of self-efficacy for symptom management immediately post intervention (Time 1) by comparing the scores from the Patient-Reported Outcomes Measurement Information System®; PROMIS® Scale. | Baseline- Week 0
  Self-efficacy for symptom management will be assessed with the PROMIS® Self Efficacy for Symptom Management Scale that contains 28 items and assess the person's current level of confidence to manage/control symptoms, manage symptoms in different settings, and keep symptoms from interfering with work, relationships, or activities. Response options are on a 5-point Likert scale (1=I am not confident at all; 5=I am very confident). Scores are summed across items, and higher scores indicate greater self-efficacy
Effects of the C-SCAT versus usual care on the primary outcomes of self-efficacy for symptom management immediately post intervention (Time 1) by comparing the scores from the Patient-Reported Outcomes Measurement Information System®; PROMIS® Scale. | 2 weeks post intervention (Timepoint 1)
  Self-efficacy for symptom management will be assessed with the PROMIS® Self Efficacy for Symptom Management Scale that contains 28 items and assess the person's current level of confidence to manage/control symptoms, manage symptoms in different settings, and keep symptoms from interfering with work, relationships, or activities. Response options are on a 5-point Likert scale (1=I am not confident at all; 5=I am very confident). Scores are summed across items, and higher scores indicate greater self-efficacy
Effects of the C-SCAT versus usual care on the primary outcomes of self-efficacy for symptom management at follow up (Time 2) by comparing the scores from the Patient-Reported Outcomes Measurement Information System®; PROMIS® Scale. | 4 weeks following Timepoint 1 (Timepoint 2)
  Self-efficacy for symptom management will be assessed with the PROMIS® Self Efficacy for Symptom Management Scale that contains 28 items and assess the person's current level of confidence to manage/control symptoms, manage symptoms in different settings, and keep symptoms from interfering with work, relationships, or activities. Response options are on a 5-point Likert scale (1=I am not confident at all; 5=I am very confident). Scores are summed across items, and higher scores indicate greater self-efficacy
Effects of the C-SCAT versus usual care on the primary outcomes of symptom self-management behaviors immediately post intervention (Time 1) by comparing the scores from the Symptom Self-management Behaviors Tool (SSMBT). | Baseline- Week 0
  The SSMBT contains 12 items with two subscales: Manage Symptoms (8 items) that addresses behaviors related to managing their symptoms, and Talk to Healthcare Provider (4 items) that addresses behaviors related to communicating with their HCP about their symptoms. Items are scored using a 5-point Likert scale (0=never/rarely; 4=always). Scores are summed across all items. Higher scores indicate higher engagement in SS-M behaviors.
Effects of the C-SCAT versus usual care on the primary outcomes of symptom self-management behaviors immediately post intervention (Time 1) by comparing the scores from the Symptom Self-management Behaviors Tool (SSMBT). | 2 weeks post intervention (Timepoint 1)
  The SSMBT contains 12 items with two subscales: Manage Symptoms (8 items) that addresses behaviors related to managing their symptoms, and Talk to Healthcare Provider (4 items) that addresses behaviors related to communicating with their HCP about their symptoms. Items are scored using a 5-point Likert scale (0=never/rarely; 4=always). Scores are summed across all items. Higher scores indicate higher engagement in SS-M behaviors.
Effects of the C-SCAT versus usual care on the primary outcomes of symptom self-management behaviors at follow up (Time 2) by comparing the scores from the Symptom Self-management Behaviors Tool (SSMBT). | 4 weeks following Timepoint 1 (Timepoint 2)
  The SSMBT contains 12 items with two subscales: Manage Symptoms (8 items) that addresses behaviors related to managing their symptoms, and Talk to Healthcare Provider (4 items) that addresses behaviors related to communicating with their HCP about their symptoms. Items are scored using a 5-point Likert scale (0=never/rarely; 4=always). Scores are summed across all items. Higher scores indicate higher engagement in SS-M behaviors.

SECONDARY OUTCOMES:
Effects of the C-SCAT versus usual care on secondary outcomes (symptom severity) at baseline, by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | Baseline-Week 0
  Symptom severity in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the severity on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (symptom severity) immediately post intervention (Time 1) by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | 2 weeks post intervention (Timepoint 1)
  Symptom severity in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the severity on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (symptom severity) immediately post intervention (Time 2) by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | 4 weeks following Timepoint 1 (Timepoint 2)
  Symptom severity in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the severity on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (symptom distress), at baseline, by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | Baseline- Week 0
  Symptom distress in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the distress on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (symptom distress) immediately post intervention (Time 1) by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | 2 weeks post intervention (Timepoint 1)
  Symptom distress in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the distress on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (symptom distress) immediately post intervention (Time 2) by comparing the scores from the Memorial Symptom Assessment Scale (MSAS). | 4 weeks following Timepoint 1 (Timepoint 2)
  Symptom distress in the past week will be assessed with the Memorial Symptom Assessment Scale (MSAS). Participants rate the distress on a 4-point Likert scale (1=slightly; 4=very severe), and the distress on a 5-point Likert scale (0=none; 4=very much).
Effects of the C-SCAT versus usual care on secondary outcomes (social function) at baseline, by comparing the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities scores. | Baseline- Week 0
  Quality of life (QOL) social function will be assessed with the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities. It contains 8 items, is scored on a 5-point Likert response scale (5=never; 1=always)
Effects of the C-SCAT versus usual care on secondary outcomes (social function) immediately post intervention (Time 1) by comparing the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities scores. | 2 weeks post intervention (Timepoint 1)
  Quality of life (QOL) social function will be assessed with the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities. It contains 8 items, is scored on a 5-point Likert response scale (5=never; 1=always)
Effects of the C-SCAT versus usual care on secondary outcomes (social function) post intervention (Time 2) by comparing the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities scores. | 4 weeks following Timepoint 1 (Timepoint 2)
  Quality of life (QOL) social function will be assessed with the PROMIS SF v2.0 Ability to Participate in Social Roles and Activities. It contains 8 items, is scored on a 5-point Likert response scale (5=never; 1=always)
Effects of the C-SCAT versus usual care on secondary outcomes (satisfaction with social function) post intervention (Time 2) by comparing the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. | Baseline -week 0
  QOL satisfaction with social function will be assessed with the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. It contains eight items, is scored on a 5-point Likert response scale (1=not at all; 5=very much)
Effects of the C-SCAT versus usual care on secondary outcomes (satisfaction with social function) post intervention (Time 2) by comparing the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. | 2 weeks post intervention (Timepoint 1)
  QOL satisfaction with social function will be assessed with the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. It contains eight items, is scored on a 5-point Likert response scale (1=not at all; 5=very much)
Effects of the C-SCAT versus usual care on secondary outcomes (satisfaction with social function) post intervention (Time 2) by comparing the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. | 4 weeks following Timepoint 1 (Timepoint 2)
  QOL satisfaction with social function will be assessed with the PROMIS SF v2.0 Satisfaction with Social Roles and Activities. It contains eight items, is scored on a 5-point Likert response scale (1=not at all; 5=very much)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Elswick, PhD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Utah Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital @ University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No